CLINICAL TRIAL: NCT01419691
Title: A Phase I Phase II Two-Step Study of the Oral Gold Compound Auranofin in Chronic Lymphocytic Leukemia (CLL)/ Small Lymphocytic Lymphoma (SLL)/ Prolymphocytic Lymphoma (PLL)
Brief Title: Phase I and II Study of Auranofin in Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: The Leukemia and Lymphoma Society (Other); Kansas Bioscience Authority (Unknown); Therapeutics for Rare and Neglected Diseases (TRND) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12838; Hem-2011-05-01 (Other Grant/Funding Number: TRND/NIH and Leukemia Lymphoma Society)
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma; Leukemia, Prolymphocytic
Keywords: auranofin; chronic lymphocytic leukemia; relapsed; refractory; CLL; SLL; PLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Recurrence | interventions — Auranofin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 2 Dose (Experimental): Auranofin 6 mg orally in the morning / 6 mg orally in the evening
  Interventions: Drug: auranofin

INTERVENTIONS:
Drug: auranofin — 6 mg twice a day for a total of 12 mg total daily dose
  Other Names: Ridaura

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of auranofin to treat patients with chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), or prolymphocytic lymphoma (PLL).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed B-cell chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), prolymphocytic leukemia arising from CLL/SLL or Richter's transformation according to WHO criteria who require therapy based on the 2008 revised IWCLL criteria.
* Relapsed or refractory disease after receiving at least 1 prior therapy for CLL
* At least 18 years old; ECOG status of 1 or less; life expectancy 2 months or greater
* Adequate organ and marrow function (total bilirubin less than 1.5x IULN; ALT less than 2x IULN; serum creatinine less than 1.5x ULN)

Exclusion Criteria:

* have had chemotherapy, radiotherapy or immunotherapy within 4 weeks prior to entering study
* have not recovered from AEs due to agents administered more than 4 weeks prior
* receiving any other investigational agent
* known second malignancy that limits survival to less than 2 years
* known HIV positive
* uncontrolled intercurrent illness
* pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Response Rate | 24 months
type, incidence, severity, seriousness and relationship to auranofin of adverse events and any laboratory abnormalities | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Suman Kambhampati, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Cancer Center, Westwood, Kansas, United States

REFERENCES:
- [Derived] Rousselle B, Massot A, Privat M, Dondaine L, Trommenschlager A, Bouyer F, Bayardon J, Ghiringhelli F, Bettaieb A, Goze C, Paul C, Malacea-Kabbara R, Bodio E. Conception and Evaluation of Fluorescent Phosphine-Gold Complexes: From Synthesis to in vivo Investigations. ChemMedChem. 2022 Jun 3;17(11):e202100773. doi: 10.1002/cmdc.202100773. Epub 2022 Mar 29. PMID 35254001